CLINICAL TRIAL: NCT05987839
Title: Early Radiographic and Clinical Outcomes of Robotic-Arm-Assisted Versus Conventional Total Knee Arthroplasty
Brief Title: Early Radiographic and Clinical Outcomes of Robotic-Arm-Assisted Versus Conventional TKA
Acronym: TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Qianfoshan Hospital (Other); Chifeng Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: robotTKARCT
Record Dates: First submitted 2023-07-19; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Total Knee Arthroplasty; Robotic

STUDY DESIGN:
Intervention Model Description: Intervention group: Total knee arthroplasty assisted by knee navigation and positioning system. Specification Model: OP-RKL22 Control group: Total knee arthroplasty without knee navigation and positioning system The same joint prosthesis was used in both the experimental group and the control group, and was approved by the manufacturer.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): Total knee arthroplasty assisted by knee navigation and positioning system. Specification Model: OP-RKL22
  Interventions: Procedure: robotic system
- control group (No Intervention): Total knee arthroplasty without knee navigation and positioning system

INTERVENTIONS:
Procedure: robotic system — Total knee arthroplasty assisted by knee navigation and positioning system
  Arms: intervention group

SUMMARY:
Purpose: A robotic system was recently introduced to improve prosthetic alignment during total knee arthroplasty (TKA). The purpose of this multicenter prospective randomized controlled trial (RCT) study was to determine whether robotic-arm-assisted TKA improves the clinical and radiological outcomes in patients compared to conventional TKA.

Methods: One hundred and thirty patients who underwent primary TKA were enrolled in this prospective, multicenter RCT conducted in 3 hospitals. Five patients were lost to follow-up at 6 weeks after surgery. Therefore, 125 patients (63 in the intervention group and 62 in the control group) remained in the final analysis. The primary outcome was the rate of patients whose mechanical axis of the femur was less than 3° deviated from the mechanical axis of the tibia evaluated by full-length weight-bearing X-rays of the lower limb at 6 weeks postoperatively. Secondary outcomes will include operation times, 6-week postoperative functional outcomes evaluated by the American Knee Society Score (KSS) and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), SF-36, adverse events (AEs) and serious adverse events (SAEs).

Hypothesis: Robotic-arm-assisted TKA is safe and effective as demonstrated in this trial.

DETAILED DESCRIPTION:
2. Materials and methods 2.1 Study design Our study was a prospective, multicenter and randomized controlled trial that was approved by the Institutional Review Board of Peking University Third Hospital (IRB # 2022-134-02), the First Affiliated Hospital of Shandong First Medical University (IRB # 2022-QX-S003-01) and Chifeng Municipal Hospital (IRB # 2022-LLSCGVK4-101-06). All patients had provided written informed consent.

2.2 Patient recruitment From November 2022 to May 2023, a total of 130 patients were randomized into two groups - 65 patients underwent robotic-assisted TKA and 65 underwent conventional TKA. The inclusion criteria were as follows: older than 18 years old and younger than 80 years old with knee osteoarthritis undergoing primary and unilateral TKA; after receiving both an oral and a written explanation of the study protocol, they provided written informed consent that they were willing to complete all of the assessments and potential interventions. The exclusion criteria were as follows: patients with infection, severe systemic disease (severe diabetes, severe osteoporosis, severe muscle loss, etc.), neuromuscular dysfunction of lower limbs, who are allergic to metal implants, participated in other clinical studies, whose knee joint has been fused for a long time without pain or deformity, unable to tolerate surgery on a systemic assessment, women who are pregnant or breastfeeding, or who expect to give birth during the clinical period, and there are other factors that affect the efficacy of observation in this study. All operations were performed by experienced surgeons for the conventional and robotic-assisted groups at three hospitals. All patients who underwent TKA with the robotic-assisted or conventional operations underwent the radiologic and clinical assessment.

Main effectiveness evaluation index The main evaluation index of the knee navigation and positioning system clinical trial was the proportion of subjects whose mechanical axis of the femoris deviated from the mechanical axis of the tibia by ≤3° on the full-length lower extremity weight-bearing X-ray at 6 weeks (±2 weeks) after surgery.

X-ray shooting requirements: Full-length weight-bearing X-ray of both lower limbs, that is, X-ray of both lower limbs including hip joint, full length of femur, knee joint, full length of tibia and fibula and ankle joint taken by the patient in the standing state. Key points: The patient stands upright on the camera frame, the back is close to the camera frame, the hands naturally droop, the knee joint is as straight as possible, the feet are the same width as the shoulders, and the internal rotation is about 15°, so that the small head of the fibula overlaps with the tibia nearly one-third, and the patella is pointed vertically in front.

The lower limb force line was evaluated by non-surgeon.

1. Measurement method of mechanical shaft of femur:

   The mechanical axis of the femur is the line from the center of the proximal joint (center of the hip joint) to the center of the distal joint (center of the knee joint).

   The central point of the hip joint is located in the central point of the femoral head circle, and the Mose circle is used to determine the central point of the femoral head. When determining the central point of the knee joint, the apex of the femoral intercondylar fossa was used as the central point of the knee joint, without measuring the width of bone tissue or soft tissue.
2. Measurement method of tibial mechanical axis:

   The mechanical axis of the tibia is the line from the center of the proximal joint (center of the knee joint) to the center of the distal joint (center of the ankle joint).

   The central point of the knee joint is located in the center of the tibial plateau. Measure the midpoint of the talus width to determine the ankle joint center point.
3. Measurement method of the medial Angle between the mechanical axis of femur and the mechanical axis of tibia:

The medial Angle between the mechanical axis of femur and the mechanical axis of tibia is the hip knee ankle Angle (HKA).

Criteria: After measurement, the Angle of HKA does not exceed 180°±3°, and it is regarded as an example of compliance with the mechanical shaft deviation Angle ≤3°. The proportion of subjects in the experimental group and the control group whose mechanical axis deviation Angle was ≤3° on the full-length lower extremity weight-bearing X-ray film 6 weeks (±2 weeks) after surgery was calculated.

Secondary effectiveness evaluation index

1. Operation time The operation time of control group was from the establishment of surgical incision to the end of skin suture. The operation start time of the experimental group was the first time when the equipment started to work and the surgical incision was established, and the operation end time was the end time of skin suture.
2. KSS score The knee society score (KSS) is one of the most commonly used scores to evaluate knee function. This method is to evaluate the patient's knee joint and its function in two aspects according to the particularity of joint replacement surgery through the evaluator interview and physical examination, that is, to obtain the information of joint anatomy, biomechanics and other aspects, and to understand the patient's functional recovery. Knee joint evaluation is to evaluate the impact of surgery on the joint and the recovery of the joint after surgery, such as: joint pain, joint range of motion, ligament stability, muscle strength, bone alignment, contracture deformity; Functional assessments include activities of daily living, walking ability, going up and down stairs, and the need for AIDS. Subjects and subjects were evaluated by KSS scale.
3. WOMAC score This score is used to assess the severity of arthritis and its therapeutic effectiveness based on the patient's relevant signs and symptoms. The structure and function of the knee joint were evaluated by pain, stiffness and joint function. The functional description of the knee joint was mainly for the lower limbs. You can use the entire system or pick a part of it when you use it. In terms of content, this rating scale assesses the structure and function of the knee joint from the three aspects of pain, stiffness, and joint function, with a total of 24 items, including the basic symptoms and signs of the entire joint. The pain part had five items, the stiffness part had two items, and the joint function part had 17 items. The reliability, validity and sensitivity of the assessment of the knee joint were objectively evaluated by the WOMAC scoring scale.
4. SF-36 Health questionnaire The SF-36 Health Survey is a universal measurement scale developed by the Medical Outcomes Study (MOS). It consists of 36 entries covering eight areas: physical function, physical role, physical pain, general health, vitality, social function, emotional role, and mental health. It is widely used in the measurement of the quality of life of the general population, the evaluation of clinical trial effect and the evaluation of health policy.

Safety evaluation

1. Incidence of adverse events Adverse events were collected and recorded throughout the clinical trial, and the incidence rate was calculated.
2. Incidence of serious adverse events Serious adverse events were collected and recorded throughout the clinical trial, and the incidence rate was calculated.

Statistical analysis and sample size calculation The description of quantitative indicators will calculate the mean, standard deviation, median, minimum, maximum, lower quartile, upper quartile, and qualitative indicators describe the frequency and frequency of each type. The comparison of two groups of general conditions will be analyzed by appropriate methods according to the type of indicators. Group t test or Wilcoxon rank sum test will be used for comparison between groups of quantitative data, U-test, chi-square test or Fisher exact probability method will be used for qualitative data, and Wilcoxon rank sum test will be used for rank data.

Test level α=0.025 (unilateral), according to β=0.2 to calculate the test grasp, the ratio of test group and control group is 1:1. According to the results of efficacy analysis, the required sample size was calculated to be 55 cases, and the sample size was expanded to 65 cases considering the 15% shedding rate. The experimental group and the control group completed 65 subjects each.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old and younger than 80 years old with knee osteoarthritis undergoing primary and unilateral TKA
* after receiving both an oral and a written explanation of the study protocol, they provided written informed consent that they were willing to complete all of the assessments and potential interventions

Exclusion Criteria:

* Allergic to metal implants
* Any active systemic and local infection
* Paralysis of muscles around the knee joint or neuropathic arthropathy
* The knee joint has been fused for a long time without pain and deformity
* Patients with severe systemic diseases (severe diabetes, severe osteoporosis, severe muscle loss, etc.), or those who cannot tolerate surgery through systemic evaluation
* Women who are pregnant or breastfeeding, or who expect to give birth during the clinical period
* Patients who are also participating in other clinical studies
* In any case, if the investigator believes that the patient is not suitable for this treatment (the patient's expectations are unrealistic or the patient has significant emotional problems)
* There are other factors that affect the efficacy of observation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
rate of alignment inlier | 6 weeks postoperatively
  the rate of patients whose mechanical axis of the femur was less than 3° deviated from the mechanical axis of the tibia evaluated by full-length weight-bearing X-rays of the lower limb at 6 weeks postoperatively

SECONDARY OUTCOMES:
operation time | Intraoperative
  The operation time of control group was from the establishment of surgical incision to the end of skin suture. The operation start time of the experimental group was the first time when the equipment started to work and the surgical incision was established, and the operation end time was the end time of skin suture.
knee society score | through study completion, an average of 6 weeks after the surgery
  The knee society score (KSS) is one of the most commonly used scores to evaluate knee function. This method is to evaluate the patient's knee joint and its function in two aspects according to the particularity of joint replacement surgery through the evaluator interview and physical examination, that is, to obtain the information of joint anatomy, biomechanics and other aspects, and to understand the patient's functional recovery. Knee joint evaluation is to evaluate the impact of surgery on the joint and the recovery of the joint after surgery, such as: joint pain, joint range of motion, ligament stability, muscle strength, bone alignment, contracture deformity; Functional assessments include activities of daily living, walking ability, going up and down stairs, and the need for AIDS. Subjects and subjects were evaluated by KSS scale. The higher the score, the better.
the Western Ontario and McMaster Universities Osteoarthritis Index | through study completion, an average of 6 weeks after the surgery
  This score is used to assess the severity of arthritis and its therapeutic effectiveness based on the patient's relevant signs and symptoms. The structure and function of the knee joint were evaluated by pain, stiffness and joint function. The functional description of the knee joint was mainly for the lower limbs. You can use the entire system or pick a part of it when you use it. In terms of content, this rating scale assesses the structure and function of the knee joint from the three aspects of pain, stiffness, and joint function, with a total of 24 items, including the basic symptoms and signs of the entire joint. The pain part had five items, the stiffness part had two items, and the joint function part had 17 items. The reliability, validity and sensitivity of the assessment of the knee joint were objectively evaluated by the Western Ontario and McMaster Universities Osteoarthritis Index. The higher the score, the better.
SF-36 | through study completion, an average of 6 weeks after the surgery
  The SF-36 Health Survey is a universal measurement scale developed by the Medical Outcomes Study (MOS). It consists of 36 entries covering eight areas: physical function, physical role, physical pain, general health, vitality, social function, emotional role, and mental health. It is widely used in the measurement of the quality of life of the general population, the evaluation of clinical trial effect and the evaluation of health policy. The higher the score, the better.
adverse events | up to 6 weeks after the surgery
  Adverse events were collected and recorded throughout the clinical trial, and the incidence rate was calculated.
serious adverse events | up to 6 weeks after the surgery
  Serious adverse events were collected and recorded throughout the clinical trial, and the incidence rate was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Yuhang, MD, Study Director — Director
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China